CLINICAL TRIAL: NCT03249896
Title: Effects of a Web/Smartphone-based Lifestyle Coaching Program on Gestational Weight Gain in Pregnant Women With Gestational Diabetes
Brief Title: Web/Smartphone-based Lifestyle Coaching Program in Pregnant Women With Gestational Diabetes
Acronym: SMART-GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Jana Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSRB 2017/00088
Record Dates: First submitted 2017-08-01; First posted 2017-08-15 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2018-11

CONDITIONS: Gestational Diabetes; Pregnancy Complications; Weight Gain
Keywords: Gestational Diabetes; RCT; Lifestyle coaching program; Smartphone app; Gestational weight gain
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications; Weight Gain; Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomised, controlled, parallel-group, single centre study. Study subjects will be randomised into either the intervention or the control arm in a 1:1 ratio. The randomisation will be stratified by ethnicity (Chinese or non-Chinese) and pre-pregnancy BMI (BMI of <25kg/m2 or ≥25kg/m2), and will be performed using computer-generated randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention arm will receive standard medical care and in addition to that, be given the Aina or Aina Mini device for self-monitoring of blood glucose (SMBG), the Habits-GDM mobile app, and a weighing scale.
  Interventions: Behavioral: Habits-GDM mobile app
- Control (No Intervention): Patients in the control arm will receive standard medical care and only be given the Aina or Aina Mini device for SMBG.
  Standard medical care involves one session of face-to-face education by a diabetes nurse educator and a dietician. Patients are initiated on capillary glucose monitoring. Subsequently, standard clinical care is provided by their obstetrician. Participation in this study will not increase the frequency of clinic visits. The frequency of SMBG will be as clinically indicated and not increased as a result of participation in this study. Should the obstetrician feels that insulin is required, it will be initiated and if necessary the patient will be referred to the endocrinology service for management of insulin therapy. In some patients, the clinician may decide to prescribe metformin.

INTERVENTIONS:
Behavioral: Habits-GDM mobile app — The intervention is a self-administered mobile app designed for GDM. It targets behavioural change by providing personalised GDM management program which consists of three main elements: lessons, tracking and coaching/feedback. Lessons contains 12 interactive modules which provide patient education on GDM. Each lesson will take approximately 10-20 minutes. Information on SMBG (linked to the Aina or Aina Mini device), weight (linked to the Bluetooth weighing scale), physical activity (physical activity tracking function in the app), and food (equipped with common local food using the Singapore food database) can be tracked and displayed visually. An interactive messaging platform is used for coaching. Generic and customised automated messages are sent from a virtual lifestyle coach to encourage and motivate patients towards healthy behaviour beneficial for GDM.
  Arms: Intervention

SUMMARY:
Gestational diabetes mellitus (GDM) affects one fifth of Singaporean pregnancies and can result in short and long term complications for mother and child. Mobile applications are effective in improving diabetes care and weight related behaviors through improved self-management. A multidisciplinary healthcare team from National University Hospital, Singapore has worked with Jana Care to develop the Habits-GDM smartphone app, a lifestyle coaching program specific for gestational diabetes. It consists of interactive lessons to provide patient education, diet, activity and weight tracking tools, messaging platform for coaching and motivating patients towards healthy behavior beneficial for gestational diabetes. It interfaces with the Aina device, a novel hardware sensor that plugs into any smartphone and can be used for glucose monitoring. This study aims to test the effectiveness of this app in preventing excessive weight gain in pregnancy among patients with gestational diabetes.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is defined as glucose intolerance of any degree with onset or first recognition during pregnancy. In Singapore, 20-30% of pregnant women are affected by GDM. If poorly controlled, GDM is associated with various maternal and perinatal morbidities such as increased cesarean deliveries, preeclampsia, preterm labour, macrosomia, neonatal hypoglycemia etc. It is well recognized now that GDM is also associated with long-term metabolic complications in mothers and offspring. Women with a history of GDM have increased risk of GDM in subsequent pregnancies, and at high risk of developing Type 2 diabetes after pregnancy. Infants born to mothers with GDM are also at increased risk of developing obesity and diabetes in later life. An increasing number of studies, including studies in Singapore, suggest that screening and management of GDM can be cost-effective, although these results are highly dependent on intervention efficacy.

In Singapore, individuals with GDM are first advised to adopt diet modification, and if glycemic control is not on target despite diet control, insulin therapy is the next line of treatment. In all cases, patients need to perform self-monitoring of blood glucose (SMBG) to guide treatment decisions. These strategies aim to reduce the risks maternal and perinatal complications. In addition to that, preventing excessive gestational weight gain (GWG) is another important goal in women with GDM. This is because excessive GWG is not only associated with higher risks of delivering a large for gestational age infant, but is also the strongest risk factor for postpartum weight retention, and an important predictor for future development of Type 2 diabetes. Lifestyle intervention programs have been shown to be effective in reducing GWG in pregnant women.

One thing in common among diet modification, SMBG and achieving optimum GWG is that they involve self-management, and hence require a certain degree of self-efficacy in women with GDM. To achieve this in the National University Hospital (NUH), patients are referred to a gestational diabetes clinic for education. At this time, if the patient's plasma glucose at 0 minute and/or 120 minutes of a 75g oral glucose tolerance test (OGTT) is <7.0 mmol/L and <11.1 mmol/L respectively, this is conducted in a group teaching session lasting 1 - 1.5 hours, with 4 - 6 patients per group, led by a diabetes nurse educator and a dietitian. If the patient's plasma glucose at 0 minutes and/or 120 minutes of a 75g OGTT is ≥7.0 and ≥11.1 mmol/L respectively, this is conducted in an individual session lasting 1 hour with a diabetes nurse educator and a dietitian. Patients are initiated on capillary glucose monitoring, typically 7 times a day, 2-3 days in a week. Subsequently, their care is provided by their obstetrician until such time as the obstetrician feels that insulin is required, in which case they are often referred back to the endocrinology service for the initiation and management of insulin therapy. Capillary glucose monitoring is carried out using a glucometer that is purchased by the patient, and the patient duly records blood glucose on a paper record which will be shown to her obstetrician at the clinic appointments every 2 - 4 weeks. In addition, weight is generally monitored at the clinic visit. Advice on diet and lifestyle modification is provided by the obstetrician based on the results of capillary glucose monitoring at the clinic visit. In between appointments, there is limited interaction between healthcare providers unless the patient identifies a problem and contacts the provider.

This arrangement has some limitations. Firstly, it has been demonstrated that spacing learning activities over a period of time improves encoding and long term retention of information. As such, the current method of providing all the education that a patient needs in a single session is less likely to be optimal for retention of information. Secondly, the collection of information (through capillary glucose monitoring) is often separated from any feedback from health care providers by days or weeks. In general, the lifestyle activities (whether diet or physical activities) which generate any abnormal blood glucose results occur in close proximity to the glucose readings (often hours before rather than weeks). By the time feedback is received, the patient often does not recall the events that generated the abnormal readings. More importantly, it does not provide any meaningful feedback to the patient that allows modification of the risk of an episode of hyperglycemia. In fact, this generates a significant amount of distress for the patient. It has been shown that the distress perceived in response to a stressor is much greater when the person experiencing the stressor does not have a way to control the occurrence of the stressor. In this context, the lack of timely feedback that is actionable related to blood glucose or weight, results in significant distress on the part of patients and results in a failure to adhere to efforts to monitor or control blood glucose. In a recent mixed-methods feasibility study to assess acceptability of mobile-application based support tool for women with GDM in NUH, most reported significant stress from the burden of management and desire for supporting tools that would aid control of blood glucose as an adjunct to self-monitoring.

It is the investigators' hypothesis that by providing education that is spaced out over 1-2 weeks and providing feedback that is timely and actionable to the patient, it will improve adherence to lifestyle modification, reduce patient distress and improve clinical outcomes for women with GDM.

Singapore has among the highest smartphone use in the world, with a smartphone adoption rate of 88%. Such widespread adoption of mobile phones and smartphone provides a promising opportunity to improve diabetes care and self-management, and to intervene on weight-related behaviors in new and exciting ways. There is emerging evidence that mobile technologies improve outcomes in patients with diabetes in the short term.

For these reasons, the investigators have developed a mobile application to aid in the management of GDM. This is carried out with a company called Jana Care. Jana Care has developed the Habits Program (http://www.habitsprogram.com), a lifestyle coaching program which is available on Apple App Store and Google Play, two of the most commonly used smartphone app platforms. This was developed based on the Diabetes Prevention Program and Look-AHEAD Trial. It targets behavioral change by providing a personalized diabetes management program which consists of 12 interactive video lessons, diet, physical activity and weight tracking tools, interactive messaging platform with the lifestyle coaches, and daily short messaging tips. It interfaces with the Aina device, a novel hardware sensor that plugs into any smartphone and can be used to measure blood glucose. The glucose readings measured are automatically transferred to the Habits Program application. It is able to generate weekly reports for patients to assess their progress.

In 2013, a pilot study was conducted by Madras Diabetes Research Foundation & Dr. Mohan's Diabetes Specialties Center, World Health Organization Collaborating Center for Non-communicable Diseases, International Diabetes Federation Center for Education, Chennai, in collaboration with Jana Care, to look at the effect of the Habits Program on changes in weight, caloric intake and physical activity in 64 overweight adults at high-risk of developing diabetes, over a period of 16 weeks. The participants achieved moderate weight loss of 4.2%, up to a maximum of 11kg. Average daily calorie and fat intake decreased by 28% and 44% respectively, while daily physical activity increased from 3438 steps (week 1) to 8459 steps (week 16) (p<0.05). Statistics collected by Jana Care from commercial deployment with approximately 13,000 individuals also showed self-reported weight loss of 4.3% and physical activity improvement of 26% at 12 weeks. Another randomized-control trial to assess the effectiveness of the program is currently underway in India, funded by the Department of Biotechnology, Government of India, in collaboration with Madras Diabetes Research Foundation, Chennai and All India Institute of Medical Sciences (AIIMS), Delhi.

The Habits Program, however, is not specifically designed for the management of GDM. Working with the Department of Obstetrics and Gynecology we have developed a workflow to manage patients with GDM by optimizing blood glucose control through lifestyle modification and achieving optimal GWG. We have worked with Jana Care to develop 'Habits-GDM' - an app modified from the Habits Program which is designed specifically to support this workflow, which takes into account the nutritional requirements and limitations on exercise during pregnancy, and the need to prevent excessive weight gain (as opposed to weight loss in the original Habits Program). The program has been customized for use in Singapore including translation (with modification of messaging) and a Singapore food database.

The investigators hypothesize that the use of a web/smartphone-based coaching program specific for the management of GDM can improve clinical outcomes among women with GDM. The investigators propose to conduct a randomised clinical trial to study the efficacy of the Habits-GDM program in clinical practice in Singapore. The primary outcome would be the percentage of patients who have excessive gestational weight gain (EGWG) according to the 2009 US Institute of Medicine (IOM) guidelines.

GDM provides an ideal clinical scenario for the use of smartphone technologies to improve self-efficacy and clinical outcomes. In Singapore, women of child bearing age well versed with using smartphone apps, these individuals are generally highly motivated, engaged to improve their own health and well-being of the fetus. In a preliminary studies, this seems to be an acceptable and preferred mode of providing information and care. The most popular option for obtaining support for management would be a web-based or smartphone app-based resource, with 58.8% of the participants rated it as their most preferred choice. More traditional source of information such as individual counselling, group teaching or printed education materials were less preferred.

Furthermore, this phase of life and intervention period is short-lived and lasts a further 5-6 months from the time of diagnosis of GDM and therefore avoids the potential problem of technology fatigue of a largely lifestyle modification intervention.

Despite pregnancy being a precious window of opportunity to bring about lasting beneficial for patients and their offspring, and smartphone-based resources being the preferred source of information by women with GDM, there are very few smartphone apps that are designed specifically to support self-management of GDM. Moreover, there is a need for such apps to be customized to the local context in terms of language, nutritional habits and food sources; and integrated to a reliable degree with existing healthcare services, clinical workflow and setup. To the investigators' knowledge, there are no such apps that fulfil these characteristics and features that are currently available in Singapore and in this region, and globally there are only two other similar trials among the GDM population which is being carried out - one in Norway and another in Ireland.

This study will result in a unique clinical application for GDM that integrates lifestyle coaching with glucose monitoring and can be used to treat GDM with minimal manpower commitment. The improved clinical outcomes are not only relevant to the current pregnancy but also have significant impact on the future metabolic health of both mothers and offspring throughout later life.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Women aged 21 years and older.
3. Singleton pregnancy.
4. GDM diagnosed between 12 to 30 weeks of gestation, based on the 2013 World Health Organization (WHO) criteria, i.e. either of the following: fasting plasma glucose ≥5.1 mmol/L, 60-minute plasma glucose ≥10.0 mmol/L, 120-minute plasma glucose ≥8.5 mmol/L, during a 75g oral glucose tolerance test (OGTT).
5. Possesses a smartphone and ability to navigate a smartphone app.
6. Proficient in English language.
7. Plan to deliver the baby in National University Hospital.

Exclusion Criteria:

1. Multiple pregnancy.
2. Pre-existing diabetes (type 1 diabetes, type 2 diabetes, or other specific types of diabetes) diagnosed prior to current pregnancy.
3. GDM diagnosed before 12 weeks of gestation.
4. No weight available in first trimester (at or before 12 weeks gestation) of the pregnancy.
5. Need for insulin therapy from the start of diagnosis of GDM, as determined by the primary clinician.
6. Heart failure.
7. Chronic kidney disease
8. Feeding and eating disorders.
9. History of bariatric surgery.
10. Long-term systemic corticosteroids use.
11. Impaired mobility.
12. Concomitant participation in another clinical study (i.e. Phase I-III clinical studies) with investigational medicinal product(s).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who have excessive gestational weight gain (EGWG) | during the pregnancy until delivery
  Percentage of patients who have EGWG is the proportion of subjects whose gestational weight gain (GWG) exceed the upper range of recommended weight gain for corresponding pre-pregnancy BMI (in this study, this is calculated using the first recorded weight and height in pregnancy at or before 12 weeks gestation) according to the 2009 IOM guidelines.
  * GWG is calculated by subtracting the first recorded weight (in kilograms) in pregnancy at or before 12 weeks gestation from the most recent weight measurement taken in the hospital (either in the clinic or in the ward) prior to delivery.
  * Pre-pregnancy BMI is calculated using the first recorded weight (in kilograms) and height (in meters) in pregnancy at or before 12 weeks gestation.

SECONDARY OUTCOMES:
Absolute GWG stratified by whether or not the subject has EGWG for the gestational weeks at recruitment | during the pregnancy until delivery
  Absolute GWG stratified by whether or not the subject has exceeded the optimal GWG for the gestational weeks at recruitment (based on the 2009 IOM guidelines).
Absolute gestational weight gain | during the pregnancy until delivery
  Absolute gestational weight gain is calculated by subtracting the first recorded weight (in kilograms) in pregnancy at or before 12 weeks gestation from the most recent weight measurement taken in the hospital (either in the clinic or in the ward) prior to delivery.
Percentage of patients who have EGWG according to the 2009 US IOM guidelines stratified by whether or not the subject has EGWG for the gestational weeks at recruitment | during the pregnancy until delivery
  Percentage of patients who have EGWG according to the 2009 US IOM guidelines stratified by whether or not the subject has exceeded the optimal GWG for the gestational weeks at recruitment
Adherence to SMBG | From recruitment until delivery
  Numbers of SMBG performed
Average readings of self-monitored blood glucose | From recruitment until delivery
  Average readings of self-monitored blood glucose
Proportion of glucose readings above glycemic targets | From recruitment until delivery
  Glycemic targets are </=5.5 mmol/L premeals, </= 6.6 mmol/L at 2 hours post meals
Proportion of subjects who progress to needing metformin and/or insulin therapy | From recruitment until delivery
  Needing metformin and/or insulin therapy in addition to diet modification
Mode of delivery | At delivery
  Vaginal delivery, assisted delivery, cesarean section
Hypertensive disorders in pregnancy | During the pregnancy until delivery
  Pregnancy induced hypertension, preeclampsia, eclampsia
Depression score | Between 35-37 weeks of gestation
  Edinburgh Postnatal Depression Scale
Anxiety score | Between 35-37 weeks of gestation
  State-Trait Anxiety Inventory
Premature delivery | At delivery
  Delivery before 37 weeks of gestation
Apgar score | At birth
  Apgar score at 1 and 5 minutes after birth
Birth weight | At birth
  Weight of the baby at birth
Shoulder dystocia | At birth
  Shoulder dystocia at birth
Birth trauma | At birth
  Birth trauma at birth
Neonatal hypoglycemia | First 24 hours from birth
  Capillary blood glucose level of <2.6mmol/L
Respiratory distress needing intubation | At birth
  Respiratory distress needing intubation
Neonatal intensive care unit admission | First 24 hours from birth
  Neonatal intensive care unit admission

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2014 Jan;37 Suppl 1:S81-90. doi: 10.2337/dc14-S081. No abstract available. PMID 24357215
- [Background] Chong YS, Cai S, Lin H, Soh SE, Lee YS, Leow MK, Chan YH, Chen L, Holbrook JD, Tan KH, Rajadurai VS, Yeo GS, Kramer MS, Saw SM, Gluckman PD, Godfrey KM, Kwek K; GUSTO study group. Ethnic differences translate to inadequacy of high-risk screening for gestational diabetes mellitus in an Asian population: a cohort study. BMC Pregnancy Childbirth. 2014 Oct 2;14:345. doi: 10.1186/1471-2393-14-345. PMID 25273851
- [Background] Yew TW, Khoo CM, Thai AC, Kale AS, Yong EL, Tai ES. The Prevalence of Gestational Diabetes Mellitus Among Asian Females is Lower Using the New 2013 World Health Organization Diagnostic Criteria. Endocr Pract. 2014 Oct;20(10):1064-9. doi: 10.4158/EP14028.OR. PMID 24936548
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Kim C, Newton KM, Knopp RH. Gestational diabetes and the incidence of type 2 diabetes: a systematic review. Diabetes Care. 2002 Oct;25(10):1862-8. doi: 10.2337/diacare.25.10.1862. PMID 12351492
- [Background] Schwartz N, Nachum Z, Green MS. The prevalence of gestational diabetes mellitus recurrence--effect of ethnicity and parity: a metaanalysis. Am J Obstet Gynecol. 2015 Sep;213(3):310-7. doi: 10.1016/j.ajog.2015.03.011. Epub 2015 Mar 7. PMID 25757637
- [Background] Catalano PM, Kirwan JP, Haugel-de Mouzon S, King J. Gestational diabetes and insulin resistance: role in short- and long-term implications for mother and fetus. J Nutr. 2003 May;133(5 Suppl 2):1674S-1683S. doi: 10.1093/jn/133.5.1674S. PMID 12730484
- [Background] Chen PY, Finkelstein EA, Ng MJ, Yap F, Yeo GS, Rajadurai VS, Chong YS, Gluckman PD, Saw SM, Kwek KY, Tan KH. Incremental Cost-Effectiveness Analysis of Gestational Diabetes Mellitus Screening Strategies in Singapore. Asia Pac J Public Health. 2016 Jan;28(1):15-25. doi: 10.1177/1010539515612908. Epub 2015 Oct 28. PMID 26512030
- [Background] Marseille E, Lohse N, Jiwani A, Hod M, Seshiah V, Yajnik CS, Arora GP, Balaji V, Henriksen O, Lieberman N, Chen R, Damm P, Metzger BE, Kahn JG. The cost-effectiveness of gestational diabetes screening including prevention of type 2 diabetes: application of a new model in India and Israel. J Matern Fetal Neonatal Med. 2013 May;26(8):802-10. doi: 10.3109/14767058.2013.765845. Epub 2013 Feb 14. PMID 23311860
- [Background] Lohse N, Marseille E, Kahn JG. Development of a model to assess the cost-effectiveness of gestational diabetes mellitus screening and lifestyle change for the prevention of type 2 diabetes mellitus. Int J Gynaecol Obstet. 2011 Nov;115 Suppl 1:S20-5. doi: 10.1016/S0020-7292(11)60007-6. PMID 22099435
- [Background] Weile LK, Kahn JG, Marseille E, Jensen DM, Damm P, Lohse N. Global cost-effectiveness of GDM screening and management: current knowledge and future needs. Best Pract Res Clin Obstet Gynaecol. 2015 Feb;29(2):206-24. doi: 10.1016/j.bpobgyn.2014.06.009. Epub 2014 Aug 21. PMID 25225056
- [Background] Goh SY, Ang SB, Bee YM, Chen YT, Gardner DS, Ho ET, Adaikan K, Lee YC, Lee CH, Lim FS, Lim HB, Lim SC, Seow J, Soh AW, Sum CF, Tai ES, Thai AC, Wong TY, Yap F. Ministry of Health Clinical Practice Guidelines: Diabetes Mellitus. Singapore Med J. 2014 Jun;55(6):334-47. doi: 10.11622/smedj.2014079. PMID 25017409
- [Background] Carreno CA, Clifton RG, Hauth JC, Myatt L, Roberts JM, Spong CY, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Sciscione A, Tolosa JE, Saade GR, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Excessive early gestational weight gain and risk of gestational diabetes mellitus in nulliparous women. Obstet Gynecol. 2012 Jun;119(6):1227-33. doi: 10.1097/AOG.0b013e318256cf1a. Erratum In: Obstet Gynecol. 2012 Sep;120(3):710. Saade, George R [added]. PMID 22617588
- [Background] Kim SY, Sharma AJ, Sappenfield W, Wilson HG, Salihu HM. Association of maternal body mass index, excessive weight gain, and gestational diabetes mellitus with large-for-gestational-age births. Obstet Gynecol. 2014 Apr;123(4):737-44. doi: 10.1097/AOG.0000000000000177. PMID 24785599
- [Background] Margerison Zilko CE, Rehkopf D, Abrams B. Association of maternal gestational weight gain with short- and long-term maternal and child health outcomes. Am J Obstet Gynecol. 2010 Jun;202(6):574.e1-8. doi: 10.1016/j.ajog.2009.12.007. Epub 2010 Feb 4. PMID 20132923
- [Background] McClure CK, Catov JM, Ness R, Bodnar LM. Associations between gestational weight gain and BMI, abdominal adiposity, and traditional measures of cardiometabolic risk in mothers 8 y postpartum. Am J Clin Nutr. 2013 Nov;98(5):1218-25. doi: 10.3945/ajcn.112.055772. Epub 2013 Sep 18. PMID 24047920
- [Background] Eades CE, Styles M, Leese GP, Cheyne H, Evans JM. Progression from gestational diabetes to type 2 diabetes in one region of Scotland: an observational follow-up study. BMC Pregnancy Childbirth. 2015 Feb 3;15:11. doi: 10.1186/s12884-015-0457-8. PMID 25643857
- [Background] Bogaerts AF, Devlieger R, Nuyts E, Witters I, Gyselaers W, Van den Bergh BR. Effects of lifestyle intervention in obese pregnant women on gestational weight gain and mental health: a randomized controlled trial. Int J Obes (Lond). 2013 Jun;37(6):814-21. doi: 10.1038/ijo.2012.162. Epub 2012 Oct 2. PMID 23032404
- [Background] Hui AL, Back L, Ludwig S, Gardiner P, Sevenhuysen G, Dean HJ, Sellers E, McGavock J, Morris M, Jiang D, Shen GX. Effects of lifestyle intervention on dietary intake, physical activity level, and gestational weight gain in pregnant women with different pre-pregnancy Body Mass Index in a randomized control trial. BMC Pregnancy Childbirth. 2014 Sep 24;14:331. doi: 10.1186/1471-2393-14-331. PMID 25248797
- [Background] Ronnberg AK, Ostlund I, Fadl H, Gottvall T, Nilsson K. Intervention during pregnancy to reduce excessive gestational weight gain-a randomised controlled trial. BJOG. 2015 Mar;122(4):537-44. doi: 10.1111/1471-0528.13131. Epub 2014 Nov 4. PMID 25367823
- [Background] Garabedian LF, Ross-Degnan D, Wharam JF. Mobile Phone and Smartphone Technologies for Diabetes Care and Self-Management. Curr Diab Rep. 2015 Dec;15(12):109. doi: 10.1007/s11892-015-0680-8. PMID 26458380
- [Background] Tufano JT, Karras BT. Mobile eHealth interventions for obesity: a timely opportunity to leverage convergence trends. J Med Internet Res. 2005 Dec 20;7(5):e58. doi: 10.2196/jmir.7.5.e58. PMID 16403722
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131
- [Background] Institute of Medicine (US) and National Research Council (US) Committee to Reexamine IOM Pregnancy Weight Guidelines; Rasmussen KM, Yaktine AL, editors. Weight Gain During Pregnancy: Reexamining the Guidelines. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32813/ PMID 20669500
- [Background] Garnweidner-Holme LM, Borgen I, Garitano I, Noll J, Lukasse M. Designing and Developing a Mobile Smartphone Application for Women with Gestational Diabetes Mellitus Followed-Up at Diabetes Outpatient Clinics in Norway. Healthcare (Basel). 2015 May 21;3(2):310-23. doi: 10.3390/healthcare3020310. PMID 27417764
- [Background] Mackillop L, Loerup L, Bartlett K, Farmer A, Gibson OJ, Hirst JE, Kenworthy Y, Kevat DA, Levy JC, Tarassenko L. Development of a real-time smartphone solution for the management of women with or at high risk of gestational diabetes. J Diabetes Sci Technol. 2014 Nov;8(6):1105-14. doi: 10.1177/1932296814542271. Epub 2014 Jul 7. PMID 25004915
- [Background] Boulos MN, Brewer AC, Karimkhani C, Buller DB, Dellavalle RP. Mobile medical and health apps: state of the art, concerns, regulatory control and certification. Online J Public Health Inform. 2014 Feb 5;5(3):229. doi: 10.5210/ojphi.v5i3.4814. eCollection 2014. PMID 24683442
- [Background] Kennelly MA, Ainscough K, Lindsay K, Gibney E, Mc Carthy M, McAuliffe FM. Pregnancy, exercise and nutrition research study with smart phone app support (Pears): Study protocol of a randomized controlled trial. Contemp Clin Trials. 2016 Jan;46:92-99. doi: 10.1016/j.cct.2015.11.018. Epub 2015 Nov 25. PMID 26625980
- [Derived] Yew TW, Chi C, Chan SY, van Dam RM, Whitton C, Lim CS, Foong PS, Fransisca W, Teoh CL, Chen J, Ho-Lim ST, Lim SL, Ong KW, Ong PH, Tai BC, Tai ES. A Randomized Controlled Trial to Evaluate the Effects of a Smartphone Application-Based Lifestyle Coaching Program on Gestational Weight Gain, Glycemic Control, and Maternal and Neonatal Outcomes in Women With Gestational Diabetes Mellitus: The SMART-GDM Study. Diabetes Care. 2021 Feb;44(2):456-463. doi: 10.2337/dc20-1216. Epub 2020 Nov 12. PMID 33184151
- See also: Consumer Barometer with Google. — http://www.consumerbarometer.com/en/graph-builder/?question=M1&filter=country:united_states,china,hong_kong_sar,korea,malaysia,singapore,australia
- See also: World Health Organization. Diagnostic criteria and classification of hyperglycaemia first detected in pregnancy. — http://www.who.int/iris/handle/10665/85975